CLINICAL TRIAL: NCT01725256
Title: A Phase 2, Multi-Center, Open-label, Randomized, Parallel-Dose Study to Determine the Safety and Efficacy of AIR001 in Subjects With WHO Group 1 Pulmonary Arterial Hypertension (PAH)
Brief Title: A Phase 2 Study to Determine the Safety and Efficacy of AIR001 in Subjects With Pulmonary Arterial Hypertension (PAH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early dt to acquisition of Sponsor and change in corporate priorities
Sponsor: Aires Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIR001-CS05
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: AIR001; sodium nitrite; PAH; Pulmonary Arterial Hypertension; inhaled sodium nitrite
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sodium Nitrite; Nitrites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 80mg AIR001 four times daily (Experimental): 80mg AIR001 nebulized four times daily for 16 weeks
  Interventions: Drug: AIR001 (sodium nitrite inhalation solution)
- 46mg AIR001 four times daily (Experimental): 46mg AIR001 nebulized four times daily for 16 weeks
  Interventions: Drug: AIR001 (sodium nitrite inhalation solution)
- 80mg AIR001 once daily (Experimental): 80mg AIR001 nebulized once daily for 16 weeks
  Interventions: Drug: AIR001 (sodium nitrite inhalation solution)

INTERVENTIONS:
Drug: AIR001 (sodium nitrite inhalation solution) — Dose arms specify dose loaded into the I-neb AAD System nebulizer
  Other Names: sodium nitrite inhalation solution; sodium nitrite; nitrite

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an investigational/experimental drug called AIR001.

To test the effectiveness, the study will evaluate how AIR001 affects the blood vessels in the lungs and the function of the heart. This will be done by monitoring changes in Pulmonary Vascular Resistance (PVR); from Baseline/Day 1 (start of study drug) to Week 16 of the study. PVR measures the resistance to flow in the blood vessels of the lungs. The study will include other assessments to evaluate the effect of the study drug on PAH, including measurements of exercise ability and evaluations of PAH disease symptoms.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of inhaled nebulized AIR001 administered, for 16 weeks, according to 3 treatment arms (80 mg once daily, 46 mg 4 times daily, or 80 mg 4 times daily) in subjects with World Health Organization (WHO) Group 1 Pulmonary Arterial Hypertension (PAH), as determined by change in Pulmonary Vascular Resistance (PVR) from Baseline to Week 16 measured immediately post completion of AIR001 nebulization (as soon as feasible).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent document
2. Able to comply with study procedures
3. Diagnosis of PAH as classified by:

   1. Idiopathic (IPAH) or heritable(HPAH); or
   2. PAH associated with CTD; Systemic Sclerosis, Limited Scleroderma, Mixed, SLE, or overlap syndrome;
   3. PAH associated with HIV ii. Simple, congenital shunts at least one year post repair. iii. Exposure to legal drugs, chemicals and toxins
4. Cardiac catheterization prior to Screening with:

   1. mPAP ≥ 25 mmHg (at rest);
   2. PCWP ≤ 15 mmHg; and
   3. PVR > 3 mmHg/L/min or 240 dyn.sec/cm5
5. A qualification cardiac catheterization, to confirm the persistence and severity of PAH, if the diagnostic catheterization was performed more than 30 days prior to Baseline

   1. Confirms diagnosis;
   2. PVR above 300 dyn.sec/cm5 to demonstrate the persistence and severity of PAH; and
   3. No change in disease-specific PAH therapy since the qualification catheterization used
6. Newly diagnosed PAH on no disease-specific PAH therapy or previously diagnosed on oral disease-specific PAH therapy for 90 days prior with either an ETRA and/or PDE-5i
7. Has PFTs within 180 days prior to Baseline with no evidence of significant parenchymal lung disease defined as:

   * FEV1 ≤ 70% (predicted) (pre-bronchodilators);
   * FEV1/FVC ≤ 70% (pre-bronchodilators); or
   * Total lung capacity < 70% (predicted).
8. Has WHO/NYHA FC II- IV.
9. ≥ 18 and ≤ 75 years.
10. Weight ≥ 40 kg.
11. Has 6MWT distance at least 50 meters.
12. Had a V/Q scan or pulmonary angiogram prior to Screening that shows no evidence of thromboembolic disease
13. If on the following: vasodilators (including calcium channel blockers), digoxin, spironolactone, or L-Arginine; must be on a stable dose 30 days prior to Baseline and maintained throughout the study
14. If on corticosteroids, has been receiving a stable dose of ≤ 20 mg/day of prednisone (or equivalent dose, if other corticosteroid) for at least 30 days
15. Women of childbearing potential must be using at least one form of medically acceptable contraception. Women who are surgically sterile or those who are post-menopausal for at least 2 years are not considered to be of childbearing potential. Men who are not sterile must also agree to use contraception

Exclusion Criteria:

1. Participation in a device or other interventional clinical studies, within 30 days of Baseline and during study participation
2. Participation in a cardio-pulmonary rehabilitation program based upon exercise within 30 days prior to Baseline and/or during the study
3. Has uncontrolled systemic hypertension: SBP > 160 millimeter of mercury (mmHg) or DBP > 100 mmHg during Screening
4. SBP < 90 mmHg at Screening or Baseline
5. History of orthostatic hypotension or at the time of Screening; defined as a drop in SBP by ≥ 20 mmHg or DBP of ≥ 10 mmHg during Screening
6. History of left-sided heart disease and/or clinically significant cardiac disease, including:

   1. Aortic or mitral valve disease (stenosis or regurgitation) defined as greater than mild;
   2. Pericardial constriction;
   3. Restrictive or congestive cardiomyopathy;
   4. Left ventricular ejection fraction < 40%
   5. Left ventricular shortening fraction < 22% by ECHO prior to Screening;
   6. Symptomatic coronary disease
7. Significant (2+ for regurgitation) valvular disease other than TR or PR
8. Acutely decompensated heart failure within 30 days prior to Baseline
9. History of atrial septostomy within 180 days prior to Baseline
10. History of obstructive sleep apnea (treated, untreated or resolved)
11. Diagnosis of Down syndrome
12. Moderate to severe hepatic impairment
13. Has chronic renal insufficiency as defined by serum creatinine > 2.5 mg/dL or has an eGFR < 30 mL/min at Screening, or requires dialysis
14. Has a Hgb concentration < 8.5 g/dL at Screening
15. Personal or family history of the following:

    1. Congenital or acquired methemoglobinemia;
    2. RBC CYPB5 reductase deficiency
16. G6PD deficiency or any contraindication to receiving methylene blue
17. For subjects with HIV any of the following:

    * Concomitant active opportunistic infections 180 days prior to Screening;
    * Detectable viral load within 90 days of Screening;
    * T-cell count < 200 mm3 within 90 days of Screening;
    * Changes in antiretroviral regimen within 90 days of Screening;
    * Using inhaled pentamidine
18. Receiving chronic treatment with prostacyclin/prostacyclin analogue within 60 days of Baseline
19. Requirement of intravenous inotropes within 30 days prior to Baseline
20. The use of oral or topical nitrates (nitroglycerin, glyceryl trinitrate (GTN), isosorbide dinitrate, and isosorbide mononitrate) within 30 days prior to Baseline and until EOS or Termination
21. Known or suspected hypersensitivity or allergic reaction to sodium nitrite or sodium nitrate
22. History of malignancy within 5-years prior to Baseline
23. Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation
24. Has a disorder that compromises the ability to give informed consent
25. Is currently pregnant or breastfeeding or intends to become pregnant
26. Investigators, study staff or their immediate families

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary vascular resistance (PVR)from baseline to week 16 assessed at peak AIR001 | 16 weeks
  The primary objective of this study is to evaluate the efficacy of inhaled nebulized AIR001 administered, for 16 weeks, according to 3 treatment arms (80 mg once daily, 46 mg 4 times daily, or 80 mg 4 times daily) in subjects with World Health Organization (WHO) Group 1 Pulmonary Arterial Hypertension (PAH), as determined by change in Pulmonary Vascular Resistance (PVR) from Baseline to Week 16 measured immediately post completion of AIR001 nebulization (as soon as feasible).

SECONDARY OUTCOMES:
Time to Clinical Worsening (TTCW), other hemodynamics, and safety | 16 weeks
  To evaluate the effect of inhaled nebulized AIR001 administered according to 3 treatment arms (80 mg once daily, 46 mg 4 times daily, or 80 mg 4 times daily) in subjects with WHO Group 1 PAH for 16 weeks, as determined by time to the first morbidity/mortality event as defined in Time to Clinical Worsening (TTCW) assessments and change from Baseline to Week 16 in the following:
  Pulmonary Vascular Resistance Index (PVRI), N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP), 6-Minute Walk Distance (6MWD) assessed at peak, 6MWD assessed prior to AIR001 nebulization (trough), Cardiac Output (CO), Cardiac Index (CI), Mean Right Atrial Pressure (mRAP), WHO/NYHA Functional Class (FC), Quality of Life (QOL) as measured by Short-Form 36 (SF-36), Borg Dyspnea Index, Mean pulmonary artery pressure (mPAP), PVR measured at trough, PVR/systemic vascular resistance (SVR) ratio at trough and peak,
  To evaluate the safety and tolerability of AIR001 in subjects with WHO Group 1 PAH.

CONTACTS AND LOCATIONS:
Overall Officials: Adaani E Frost, M.D., Principal Investigator — Baylor College of Medicine
Locations (25):
- United States (17):
  - UCSD Medical Center, La Jolla, California
  - UCLA Medical Center, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (4):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Alfred Hospital, Melbourne, Victoria
- Hungary (4):
  - Gottsegen Gyorgy Hungarian, Budapest
  - Semmelweis Karlocai, Budapest
  - University of Debrecen, Debrecen
  - University of Szeged, Szeged

REFERENCES:
- [Background] Ahanchi SS, Tsihlis ND, Kibbe MR. The role of nitric oxide in the pathophysiology of intimal hyperplasia. J Vasc Surg. 2007 Jun;45 Suppl A:A64-73. doi: 10.1016/j.jvs.2007.02.027. PMID 17544026
- [Background] Alef MJ, Vallabhaneni R, Carchman E, Morris SM Jr, Shiva S, Wang Y, Kelley EE, Tarpey MM, Gladwin MT, Tzeng E, Zuckerbraun BS. Nitrite-generated NO circumvents dysregulated arginine/NOS signaling to protect against intimal hyperplasia in Sprague-Dawley rats. J Clin Invest. 2011 Apr;121(4):1646-56. doi: 10.1172/JCI44079. Epub 2011 Mar 23. PMID 21436585
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Badesch DB, Champion HC, Gomez Sanchez MA, Hoeper MM, Loyd JE, Manes A, McGoon M, Naeije R, Olschewski H, Oudiz RJ, Torbicki A. Diagnosis and assessment of pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S55-S66. doi: 10.1016/j.jacc.2009.04.011. PMID 19555859
- [Background] Bailey SJ, Winyard P, Vanhatalo A, Blackwell JR, Dimenna FJ, Wilkerson DP, Tarr J, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of low-intensity exercise and enhances tolerance to high-intensity exercise in humans. J Appl Physiol (1985). 2009 Oct;107(4):1144-55. doi: 10.1152/japplphysiol.00722.2009. Epub 2009 Aug 6. PMID 19661447
- [Background] Barbosa PB, Ferreira EM, Arakaki JS, Takara LS, Moura J, Nascimento RB, Nery LE, Neder JA. Kinetics of skeletal muscle O2 delivery and utilization at the onset of heavy-intensity exercise in pulmonary arterial hypertension. Eur J Appl Physiol. 2011 Aug;111(8):1851-61. doi: 10.1007/s00421-010-1799-6. Epub 2011 Jan 12. PMID 21225278
- [Background] Battistini B, Berthiaume N, Kelland NF, Webb DJ, Kohan DE. Profile of past and current clinical trials involving endothelin receptor antagonists: the novel "-sentan" class of drug. Exp Biol Med (Maywood). 2006 Jun;231(6):653-95. PMID 16740981
- [Background] Battle RW, Davitt MA, Cooper SM, Buckley LM, Leib ES, Beglin PA, Tischler MD. Prevalence of pulmonary hypertension in limited and diffuse scleroderma. Chest. 1996 Dec;110(6):1515-9. doi: 10.1378/chest.110.6.1515. PMID 8989070
- [Background] Bergstra A, van den Heuvel AF, Zijlstra F, Berger RM, Mook GA, van Veldhuisen DJ. Validation of Fick cardiac output calculated with assumed oxygen consumption: a study of cardiac output during epoprostenol. Neth Heart J. 2004 May;12(5):208-213. PMID 25696328
- [Background] Channick RN, Olschewski H, Seeger W, Staub T, Voswinckel R, Rubin LJ. Safety and efficacy of inhaled treprostinil as add-on therapy to bosentan in pulmonary arterial hypertension. J Am Coll Cardiol. 2006 Oct 3;48(7):1433-7. doi: 10.1016/j.jacc.2006.05.070. Epub 2006 Sep 14. PMID 17010807
- [Background] Chaouat A, Bugnet AS, Kadaoui N, Schott R, Enache I, Ducolone A, Ehrhart M, Kessler R, Weitzenblum E. Severe pulmonary hypertension and chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Jul 15;172(2):189-94. doi: 10.1164/rccm.200401-006OC. Epub 2005 Apr 14. PMID 15831842
- [Background] Clozel M, Breu V, Gray GA, Kalina B, Loffler BM, Burri K, Cassal JM, Hirth G, Muller M, Neidhart W, et al. Pharmacological characterization of bosentan, a new potent orally active nonpeptide endothelin receptor antagonist. J Pharmacol Exp Ther. 1994 Jul;270(1):228-35. PMID 8035319
- [Background] Cosby K, Partovi KS, Crawford JH, Patel RP, Reiter CD, Martyr S, Yang BK, Waclawiw MA, Zalos G, Xu X, Huang KT, Shields H, Kim-Shapiro DB, Schechter AN, Cannon RO 3rd, Gladwin MT. Nitrite reduction to nitric oxide by deoxyhemoglobin vasodilates the human circulation. Nat Med. 2003 Dec;9(12):1498-505. doi: 10.1038/nm954. Epub 2003 Nov 2. PMID 14595407
- [Background] Dejam A, Hunter CJ, Tremonti C, Pluta RM, Hon YY, Grimes G, Partovi K, Pelletier MM, Oldfield EH, Cannon RO 3rd, Schechter AN, Gladwin MT. Nitrite infusion in humans and nonhuman primates: endocrine effects, pharmacokinetics, and tolerance formation. Circulation. 2007 Oct 16;116(16):1821-31. doi: 10.1161/CIRCULATIONAHA.107.712133. Epub 2007 Sep 24. PMID 17893272
- [Background] Farber HW, Loscalzo J. Pulmonary arterial hypertension. N Engl J Med. 2004 Oct 14;351(16):1655-65. doi: 10.1056/NEJMra035488. No abstract available. PMID 15483284
- [Background] Task Force for Diagnosis and Treatment of Pulmonary Hypertension of European Society of Cardiology (ESC); European Respiratory Society (ERS); International Society of Heart and Lung Transplantation (ISHLT); Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G. Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Respir J. 2009 Dec;34(6):1219-63. doi: 10.1183/09031936.00139009. Epub 2009 Sep 12. No abstract available. PMID 19749199
- [Background] Ghofrani HA, Barst RJ, Benza RL, Champion HC, Fagan KA, Grimminger F, Humbert M, Simonneau G, Stewart DJ, Ventura C, Rubin LJ. Future perspectives for the treatment of pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S108-S117. doi: 10.1016/j.jacc.2009.04.014. PMID 19555854
- [Background] Giaid A, Saleh D. Reduced expression of endothelial nitric oxide synthase in the lungs of patients with pulmonary hypertension. N Engl J Med. 1995 Jul 27;333(4):214-21. doi: 10.1056/NEJM199507273330403. PMID 7540722
- [Background] Gielis JF, Lin JY, Wingler K, Van Schil PE, Schmidt HH, Moens AL. Pathogenetic role of eNOS uncoupling in cardiopulmonary disorders. Free Radic Biol Med. 2011 Apr 1;50(7):765-76. doi: 10.1016/j.freeradbiomed.2010.12.018. Epub 2010 Dec 21. PMID 21172428
- [Background] Gladwin MT, Raat NJ, Shiva S, Dezfulian C, Hogg N, Kim-Shapiro DB, Patel RP. Nitrite as a vascular endocrine nitric oxide reservoir that contributes to hypoxic signaling, cytoprotection, and vasodilation. Am J Physiol Heart Circ Physiol. 2006 Nov;291(5):H2026-35. doi: 10.1152/ajpheart.00407.2006. Epub 2006 Jun 23. PMID 16798825
- [Background] Gladwin MT, Vichinsky E. Pulmonary complications of sickle cell disease. N Engl J Med. 2008 Nov 20;359(21):2254-65. doi: 10.1056/NEJMra0804411. No abstract available. PMID 19020327
- [Background] Hassoun PM, Mouthon L, Barbera JA, Eddahibi S, Flores SC, Grimminger F, Jones PL, Maitland ML, Michelakis ED, Morrell NW, Newman JH, Rabinovitch M, Schermuly R, Stenmark KR, Voelkel NF, Yuan JX, Humbert M. Inflammation, growth factors, and pulmonary vascular remodeling. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S10-S19. doi: 10.1016/j.jacc.2009.04.006. PMID 19555853
- [Background] Hassoun PM. Pulmonary arterial hypertension complicating connective tissue disease. In: Humbert, M, Lynch JP, Eds. Pulmonary Hypertension. New York: Informa Healthcare USA, Inc. 2010: 161-175
- [Background] Humbert M, Morrell NW, Archer SL, Stenmark KR, MacLean MR, Lang IM, Christman BW, Weir EK, Eickelberg O, Voelkel NF, Rabinovitch M. Cellular and molecular pathobiology of pulmonary arterial hypertension. J Am Coll Cardiol. 2004 Jun 16;43(12 Suppl S):13S-24S. doi: 10.1016/j.jacc.2004.02.029. PMID 15194174
- [Background] Humbert M, Sitbon O, Simonneau G. Treatment of pulmonary arterial hypertension. N Engl J Med. 2004 Sep 30;351(14):1425-36. doi: 10.1056/NEJMra040291. No abstract available. PMID 15459304
- [Background] Hunter CJ, Dejam A, Blood AB, Shields H, Kim-Shapiro DB, Machado RF, Tarekegn S, Mulla N, Hopper AO, Schechter AN, Power GG, Gladwin MT. Inhaled nebulized nitrite is a hypoxia-sensitive NO-dependent selective pulmonary vasodilator. Nat Med. 2004 Oct;10(10):1122-7. doi: 10.1038/nm1109. Epub 2004 Sep 12. PMID 15361865
- [Background] Kiowski W, Sutsch G, Hunziker P, Muller P, Kim J, Oechslin E, Schmitt R, Jones R, Bertel O. Evidence for endothelin-1-mediated vasoconstriction in severe chronic heart failure. Lancet. 1995 Sep 16;346(8977):732-6. doi: 10.1016/s0140-6736(95)91504-4. PMID 7658874
- [Background] Krowka MJ, Swanson KL, Frantz RP, McGoon MD, Wiesner RH. Portopulmonary hypertension: Results from a 10-year screening algorithm. Hepatology. 2006 Dec;44(6):1502-10. doi: 10.1002/hep.21431. PMID 17133488
- [Background] Lansley KE, Winyard PG, Bailey SJ, Vanhatalo A, Wilkerson DP, Blackwell JR, Gilchrist M, Benjamin N, Jones AM. Acute dietary nitrate supplementation improves cycling time trial performance. Med Sci Sports Exerc. 2011 Jun;43(6):1125-31. doi: 10.1249/MSS.0b013e31821597b4. PMID 21471821
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Effects of dietary nitrate on oxygen cost during exercise. Acta Physiol (Oxf). 2007 Sep;191(1):59-66. doi: 10.1111/j.1748-1716.2007.01713.x. Epub 2007 Jul 17. PMID 17635415
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Dietary nitrate reduces maximal oxygen consumption while maintaining work performance in maximal exercise. Free Radic Biol Med. 2010 Jan 15;48(2):342-7. doi: 10.1016/j.freeradbiomed.2009.11.006. Epub 2009 Nov 12. PMID 19913611
- [Background] Larsen FJ, Schiffer TA, Borniquel S, Sahlin K, Ekblom B, Lundberg JO, Weitzberg E. Dietary inorganic nitrate improves mitochondrial efficiency in humans. Cell Metab. 2011 Feb 2;13(2):149-59. doi: 10.1016/j.cmet.2011.01.004. PMID 21284982
- [Background] Levi, DS, Scott V, et al. Pulmonary arterial hypertension in congenital heart disease. In: Humbert, M, Lynch, JP, Eds. Pulmonary Hypertension. New York: Informa Healthcare USA, Inc. 2010: 176-195.
- [Background] Mainguy V, Maltais F, Saey D, Gagnon P, Martel S, Simon M, Provencher S. Peripheral muscle dysfunction in idiopathic pulmonary arterial hypertension. Thorax. 2010 Feb;65(2):113-7. doi: 10.1136/thx.2009.117168. Epub 2009 Aug 30. PMID 19720606
- [Background] McLaughlin VV, Archer SL, Badesch DB, Barst RJ, Farber HW, Lindner JR, Mathier MA, McGoon MD, Park MH, Rosenson RS, Rubin LJ, Tapson VF, Varga J; American College of Cardiology Foundation Task Force on Expert Consensus Documents; American Heart Association; American College of Chest Physicians; American Thoracic Society, Inc; Pulmonary Hypertension Association. ACCF/AHA 2009 expert consensus document on pulmonary hypertension a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents and the American Heart Association developed in collaboration with the American College of Chest Physicians; American Thoracic Society, Inc.; and the Pulmonary Hypertension Association. J Am Coll Cardiol. 2009 Apr 28;53(17):1573-619. doi: 10.1016/j.jacc.2009.01.004. No abstract available. PMID 19389575
- [Background] Mehta NJ, Khan IA, Mehta RN, Sepkowitz DA. HIV-Related pulmonary hypertension: analytic review of 131 cases. Chest. 2000 Oct;118(4):1133-41. doi: 10.1378/chest.118.4.1133. PMID 11035689
- [Background] Morrell NW, Adnot S, Archer SL, Dupuis J, Lloyd Jones P, MacLean MR, McMurtry IF, Stenmark KR, Thistlethwaite PA, Weissmann N, Yuan JX, Weir EK. Cellular and molecular basis of pulmonary arterial hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S20-S31. doi: 10.1016/j.jacc.2009.04.018. PMID 19555855
- [Background] Mukerjee D, St George D, Coleiro B, Knight C, Denton CP, Davar J, Black CM, Coghlan JG. Prevalence and outcome in systemic sclerosis associated pulmonary arterial hypertension: application of a registry approach. Ann Rheum Dis. 2003 Nov;62(11):1088-93. doi: 10.1136/ard.62.11.1088. PMID 14583573
- [Background] Olschewski H, Rohde B, Behr J, Ewert R, Gessler T, Ghofrani HA, Schmehl T. Pharmacodynamics and pharmacokinetics of inhaled iloprost, aerosolized by three different devices, in severe pulmonary hypertension. Chest. 2003 Oct;124(4):1294-304. doi: 10.1378/chest.124.4.1294. PMID 14555558
- [Background] Opravil M, Pechere M, Speich R, Joller-Jemelka HI, Jenni R, Russi EW, Hirschel B, Luthy R. HIV-associated primary pulmonary hypertension. A case control study. Swiss HIV Cohort Study. Am J Respir Crit Care Med. 1997 Mar;155(3):990-5. doi: 10.1164/ajrccm.155.3.9117037.
- [Background] Piazza G, Goldhaber SZ. Chronic thromboembolic pulmonary hypertension. N Engl J Med. 2011 Jan 27;364(4):351-60. doi: 10.1056/NEJMra0910203. No abstract available. PMID 21268727
- [Background] Pluta RM, Dejam A, Grimes G, Gladwin MT, Oldfield EH. Nitrite infusions to prevent delayed cerebral vasospasm in a primate model of subarachnoid hemorrhage. JAMA. 2005 Mar 23;293(12):1477-84. doi: 10.1001/jama.293.12.1477. PMID 15784871
- [Background] Pluta RM, Oldfield EH, Bakhtian KD, Fathi AR, Smith RK, Devroom HL, Nahavandi M, Woo S, Figg WD, Lonser RR. Safety and feasibility of long-term intravenous sodium nitrite infusion in healthy volunteers. PLoS One. 2011 Jan 10;6(1):e14504. doi: 10.1371/journal.pone.0014504. PMID 21249218
- [Background] Ranque B, Authier FJ, Berezne A, Guillevin L, Mouthon L. Systemic sclerosis-associated myopathy. Ann N Y Acad Sci. 2007 Jun;1108:268-82. doi: 10.1196/annals.1422.029. PMID 17899625
- [Background] Rubin LJ. Primary pulmonary hypertension. N Engl J Med. 1997 Jan 9;336(2):111-7. doi: 10.1056/NEJM199701093360207. No abstract available. PMID 8988890
- [Background] Rubin LJ; American College of Chest Physicians. Diagnosis and management of pulmonary arterial hypertension: ACCP evidence-based clinical practice guidelines. Chest. 2004 Jul;126(1 Suppl):7S-10S. doi: 10.1378/chest.126.1_suppl.7S. No abstract available. PMID 15249491
- [Background] Shiva S. Mitochondria as metabolizers and targets of nitrite. Nitric Oxide. 2010 Feb 15;22(2):64-74. doi: 10.1016/j.niox.2009.09.002. Epub 2009 Sep 27. PMID 19788924
- [Background] Shorr AF, Helman DL, Davies DB, Nathan SD. Pulmonary hypertension in advanced sarcoidosis: epidemiology and clinical characteristics. Eur Respir J. 2005 May;25(5):783-8. doi: 10.1183/09031936.05.00083404. PMID 15863633
- [Background] Simonneau G, Robbins IM, Beghetti M, Channick RN, Delcroix M, Denton CP, Elliott CG, Gaine SP, Gladwin MT, Jing ZC, Krowka MJ, Langleben D, Nakanishi N, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2009 Jun 30;54(1 Suppl):S43-S54. doi: 10.1016/j.jacc.2009.04.012. PMID 19555858
- [Background] Sitbon O, Lascoux-Combe C, Delfraissy JF, Yeni PG, Raffi F, De Zuttere D, Gressin V, Clerson P, Sereni D, Simonneau G. Prevalence of HIV-related pulmonary arterial hypertension in the current antiretroviral therapy era. Am J Respir Crit Care Med. 2008 Jan 1;177(1):108-13. doi: 10.1164/rccm.200704-541OC. Epub 2007 Oct 11. PMID 17932378
- [Background] Smith AP, Demoncheaux EA, Higenbottam TW. Nitric oxide gas decreases endothelin-1 mRNA in cultured pulmonary artery endothelial cells. Nitric Oxide. 2002 Mar;6(2):153-9. doi: 10.1006/niox.2001.0400. PMID 11890739
- [Background] Souza R, Humbert M, Sztrymf B, Jais X, Yaici A, Le Pavec J, Parent F, Herve P, Soubrier F, Sitbon O, Simonneau G. Pulmonary arterial hypertension associated with fenfluramine exposure: report of 109 cases. Eur Respir J. 2008 Feb;31(2):343-8. doi: 10.1183/09031936.00104807. Epub 2007 Oct 24. PMID 17959632
- [Background] Tsihlis ND, Oustwani CS, Vavra AK, Jiang Q, Keefer LK, Kibbe MR. Nitric oxide inhibits vascular smooth muscle cell proliferation and neointimal hyperplasia by increasing the ubiquitination and degradation of UbcH10. Cell Biochem Biophys. 2011 Jun;60(1-2):89-97. doi: 10.1007/s12013-011-9179-3. PMID 21448667
- [Background] Tyvaso US Package Insert. Research Triangle Park, NC: United Therapeutics Corp; 2011.
- [Background] Uhlmann D, Ludwig S, Escher E, Armann B, Gabel G, Teupser D, Tannapfel A, Hauss J, Witzigmann H. Protective effect of a selective endothelin a receptor antagonist (BSF 208075) on graft pancreatitis in pig pancreas transplantation. Transplant Proc. 2001 Nov-Dec;33(7-8):3732-4. doi: 10.1016/s0041-1345(01)02523-4. No abstract available. PMID 11750590
- [Background] Vanhatalo A, Fulford J, Bailey SJ, Blackwell JR, Winyard PG, Jones AM. Dietary nitrate reduces muscle metabolic perturbation and improves exercise tolerance in hypoxia. J Physiol. 2011 Nov 15;589(Pt 22):5517-28. doi: 10.1113/jphysiol.2011.216341. Epub 2011 Sep 12. PMID 21911616
- [Background] Voswinckel R, Enke B, Reichenberger F, Kohstall M, Kreckel A, Krick S, Gall H, Gessler T, Schmehl T, Ghofrani HA, Schermuly RT, Grimminger F, Rubin LJ, Seeger W, Olschewski H. Favorable effects of inhaled treprostinil in severe pulmonary hypertension: results from randomized controlled pilot studies. J Am Coll Cardiol. 2006 Oct 17;48(8):1672-81. doi: 10.1016/j.jacc.2006.06.062. Epub 2006 Sep 26. PMID 17045906
- [Background] Ware, JE, Kosinski, M, Dewey JE. How to Score Version Two of the SF-36 Health Survey. Lincoln, RI: QualityMetric, Incorporated, 2000.
- [Background] Weber C, Schmitt R, Birnboeck H, Hopfgartner G, van Marle SP, Peeters PA, Jonkman JH, Jones CR. Pharmacokinetics and pharmacodynamics of the endothelin-receptor antagonist bosentan in healthy human subjects. Clin Pharmacol Ther. 1996 Aug;60(2):124-37. doi: 10.1016/S0009-9236(96)90127-7. PMID 8823230
- [Background] Weitzenblum E, Chaouat A. Severe pulmonary hypertension in COPD: is it a distinct disease? Chest. 2005 May;127(5):1480-2. doi: 10.1378/chest.127.5.1480. No abstract available. PMID 15888814
- [Background] Williamson DJ, Wallman LL, Jones R, Keogh AM, Scroope F, Penny R, Weber C, Macdonald PS. Hemodynamic effects of Bosentan, an endothelin receptor antagonist, in patients with pulmonary hypertension. Circulation. 2000 Jul 25;102(4):411-8. doi: 10.1161/01.cir.102.4.411. PMID 10908213
- [Background] Zuckerbraun BS, George P, Gladwin MT. Nitrite in pulmonary arterial hypertension: therapeutic avenues in the setting of dysregulated arginine/nitric oxide synthase signalling. Cardiovasc Res. 2011 Feb 15;89(3):542-52. doi: 10.1093/cvr/cvq370. Epub 2010 Dec 22. PMID 21177703